CLINICAL TRIAL: NCT07024875
Title: Precision Neuroimaging of Parkinson's Disease
Brief Title: Neuroimaging of Parkinson's
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202410006; R01NS140256 (NIH)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Parkinsons Disease (PD)
Keywords: Neurology; Radiology; FMRI; Precision Neuroimaging; Resting-State Functional Connectivity; Subcortical Structures; Functional MRI; Brain Imaging Data Structure; Gait Analysis; Motor Cortex Connectivity; Non-Demented Parkinson's; Openneuro Repository; Observational Cohort Study; Action Initiation; Freezing of Gait; Parkinson's Disease; Somato-Cognitive Action Network (SCAN); Precision Functional Mapping; Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Participants: * 70 non-demented individuals with clinically definite PD
  * Must be 40 years of age or older
  * Both male & female
- Healthy Control: * 50 individuals with normal neurological exams and cognition
  * No first-degree relatives with PD
  * Also, must be 40 years of age or older

SUMMARY:
Parkinson's Disease (PD) is a neurodegenerative disorder caused by dysfunction in both subcortical structures and the cortex. The investigators recently discovered a new brain system called the Somato-Cognitive Action Network (SCAN), which could be a primary locus of dysfunction in PD. Here, the investigators will use magnetic resonance imaging techniques in PD patients to test whether SCAN is critical for PD. The investigators will determine whether SCAN is connected to PD-relevant subcortical structures, and whether PD patients exhibit altered subcortical-to-SCAN connectivity. If successful, this work will identify SCAN as a specific circuit altered in PD patients that can serve as a new target for future neuromodulatory PD therapies.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neurodegenerative disease that causes symptoms such as tremor, bradykinesia, and freezing of gait, as well as sleep disturbance, autonomic dysfunction, and abulia. PD patients particularly struggle to initiate and maintain actions, which causes gait freezing, leading to falls. PD results from dysfunction in motor circuitry, including connections between subcortical structures such as substantia nigra and striatum, as well as primary motor cortex, which drives voluntary movement.

Recently, our group rewrote the textbook diagrams of motor circuitry. The investigators described a previously unrecognized Somato-Cognitive Action Network (SCAN) which is interspersed between effector-specific regions of primary motor cortex (foot, hand, mouth). The SCAN is engaged by coordinated rather than isolated actions, and it is strongly preferentially connected to other cortical regions important for action planning and control, autonomic function, and arousal.

Many SCAN functions (drive to act, gait, autonomic control, arousal, motor coordination) are affected in PD. Further, clinical targets for neuromodulation in PD are connected to SCAN. Thus, SCAN dysfunction might be an important aspect of PD pathophysiology and resulting symptoms. Critically, recent technical advances in noninvasive functional neuroimaging allow us for the first time to reliably evaluate the connectivity of motor systems, including SCAN, into the deep subcortical structures most relevant for PD.

Using these patient-oriented techniques, the investigators will first test whether PD-relevant subcortical structures-including clinical targets for PD-are connected more strongly to the SCAN circuit than to effector-specific M1 foot, hand, and mouth regions. The investigators will then test whether these subcortical-to-SCAN circuits are altered in PD patients to a greater degree than effector-specific circuits.

This work will advance a new conceptualization of PD as a disorder of SCAN rather than of traditional effector-specific M1, which will revolutionize how the investigators think of the disorder. Localizing PD disruption to specific portions of M1 could aid with evaluation of patients using these advanced, noninvasive fMRI techniques, and can provide precision targets of interest for other imaging modalities. Noninvasive mapping of cortico-subcortical connectivity will enable optimal target definition for neuromodulatory treatment of PD. Reconceptualizing PD as a disorder of SCAN, a system for integrated action, rather than of M1 circuits for isolated movement, may spur development of alternate symptom evaluation tools oriented around this framework. Finally, localizing M1 sites of disruption in PD opens the possibility of treating PD using cortical stimulation, a less-invasive alternative to deep brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Must meet specific health and cognitive criteria depending on the group. For PD participants
* Clinical diagnosis of Parkinson's Disease
* Must not meet dementia criteria For Healthy Control Participants
* Normal or benign neurological exam
* Normal cognition
* No first-degree relatives with Parkinson's Disease

Exclusion Criteria:

1. Neurological Disorders (other than PD)

   - Any other neurological condition
2. Significant Head Injury

   * Head injury with loss of consciousness >5 minutes
   * Or any neurological sequelae
3. Psychiatric Disorders

   * Schizophrenia
   * Bipolar Disorder
   * Epilepsy
4. Serious Medical Conditions

   * End-stage organ failure
   * Ongoing cancer treatment
5. Cognitive Impairment

   * Diagnosis of dementia
   * MMSE score <24 or MoCA score <21
6. MRI contraindications

   * Metal implants
   * claustrophobia
   * Weight over 300 lbs (due to weight restrictions of the MRI scanner)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Parkinson's Disease (PD) Patients
     * 70 non-demented individuals with clinically definite PD
     * Must be 50 years of age or older
     * Both male & female
     * Must not meet dementia criteria
  2. Age-matched Healthy Controls
     * 50 individuals with normal neurological exams and cognition
     * No first degree relatives with PD
     * Also, must be 50 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Cortico-subcortical connectivity to SCAN vs effectors | 3 months per participant, across three 2-hour MRI scan sessions.
  We will collect resting-state functional magnetic resonance imaging (fMRI) scans from the brains of all participants. From the fMRI scans, we will compute the functional connectivity between each of the subcortical brain structures relevant for Parkinson's disease (including substantia nigra, subthalamic nucleus, globus pallidus internus, and ventral intermediate nucleus of the thalamus) and each subdivision of primary motor cortex (Somato-Cognitive Action network and effector-specific regions controlling the hand, foot, and face). Functional connectivity will be computed as pairwise temporal correlations of the activity timecourses in each location.
  We hypothesize that subcortical structures will exhibit differential functional connectivity to the Somato-Cognitive Action network than to the effector-specific regions of primary motor cortex.

SECONDARY OUTCOMES:
Cortico-subcortical connectivity to SCAN in Parkinson's and controls | 3 months per participant, across three 2-hour MRI scan sessions.
  We will collect resting-state functional magnetic resonance imaging (fMRI) scans from the brains of all participants. From the fMRI scans, we will compute the functional connectivity between each of the subcortical brain structures relevant for Parkinson's disease (including substantia nigra, subthalamic nucleus, globus pallidus internus, and ventral intermediate nucleus of the thalamus) and each subdivision of primary motor cortex (Somato-Cognitive Action network and effector-specific regions controlling the hand, foot, and face). Functional connectivity will be computed as pairwise temporal correlations of the activity timecourses in each location.
  We hypothesize that people with Parkinson's Disease will exhibit differential functional connectivity than controls between subcortical structures and the Somato-Cognitive Action network.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Gordon, PhD, Principal Investigator — Washington University School of Medicine; Nico Dosenbach, MD/PhD, Principal Investigator — Washington University School of Medicine; Scott Norris, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- East Imaging Building, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD, including de-identified neuroimaging data, summary measures from clinical and motor assessments, summary measures from behavioral tasks, summary measures from psychiatric questionnaires, & anonymized demographic data.
Supporting Information: Analytic Code
Time Frame: IPD and supporting information will be available after initial publication and shared indefinitely.
Access Criteria: IPD and supporting information will be publicly accessible through the OpenNeuro repository (https://openneuro.org). Openneuro provides a persistent unique Accession Number for deposited datasets. All publications associated with this data will reference that Accession Number.

REFERENCES:
- [Background] Cui W, Wang Y, Ren J, Hubbard CS, Fu X, Fang S, Wang D, Zhang H, Li Y, Li L, Jiang T, Liu H. Personalized fMRI Delineates Functional Regions Preserved within Brain Tumors. Ann Neurol. 2022 Mar;91(3):353-366. doi: 10.1002/ana.26303. Epub 2022 Jan 31. PMID 35023218
- [Background] Ren J, Chi Q, Hubbard CS, Cui W, Wang D, Li L, Zhang H, Liu H. Personalized functional imaging identifies brain stimulation target for a patient with trauma-induced functional disruption. Brain Stimul. 2022 Jan-Feb;15(1):53-56. doi: 10.1016/j.brs.2021.11.005. Epub 2021 Nov 5. No abstract available. PMID 34749006
- [Background] Guo Y, Ren J, Cui W, Dahmani L, Wang D, Fu X, Li M, Li S, Zhang Y, Lin X, Zhen Z, Xu Y, Xie D, Guan H, Yi F, Wang J, Shi Q, Liu H. Personalized brain MRI revealed distinct functional and anatomical disruptions in Creutzfeldt-Jakob disease and Alzheimer's disease. CNS Neurosci Ther. 2024 Feb;30(2):e14404. doi: 10.1111/cns.14404. Epub 2023 Aug 14. PMID 37577861
- [Background] Dahmani L, Bai Y, Li M, Ren J, Shen L, Ma J, Li H, Wei W, Li P, Wang D, Du L, Cui W, Liu H, Wang M. Focused ultrasound thalamotomy for tremor treatment impacts the cerebello-thalamo-cortical network. NPJ Parkinsons Dis. 2023 Jun 15;9(1):90. doi: 10.1038/s41531-023-00543-8. PMID 37322044
- [Background] Ji GJ, Liu T, Li Y, Liu P, Sun J, Chen X, Tian Y, Chen X, Dahmani L, Liu H, Wang K, Hu P. Structural correlates underlying accelerated magnetic stimulation in Parkinson's disease. Hum Brain Mapp. 2021 Apr 15;42(6):1670-1681. doi: 10.1002/hbm.25319. Epub 2020 Dec 14. PMID 33314545
- [Background] Hill KK, Campbell MC, McNeely ME, Karimi M, Ushe M, Tabbal SD, Hershey T, Flores HP, Hartlein JM, Lugar HM, Revilla FJ, Videen TO, Earhart GM, Perlmutter JS. Cerebral blood flow responses to dorsal and ventral STN DBS correlate with gait and balance responses in Parkinson's disease. Exp Neurol. 2013 Mar;241:105-12. doi: 10.1016/j.expneurol.2012.12.003. Epub 2012 Dec 19. PMID 23262122
- [Background] Myers PS, McNeely ME, Koller JM, Earhart GM, Campbell MC. Cerebellar Volume and Executive Function in Parkinson Disease with and without Freezing of Gait. J Parkinsons Dis. 2017;7(1):149-157. doi: 10.3233/JPD-161029. PMID 28106569
- [Background] Horin AP, Myers PS, Pickett KA, Earhart GM, Campbell MC. Resting-state functional connectivity associated with gait characteristics in people with Parkinson's disease. Behav Brain Res. 2021 Aug 6;411:113398. doi: 10.1016/j.bbr.2021.113398. Epub 2021 Jun 2. PMID 34087255
- [Background] Maiti B, Rawson KS, Tanenbaum AB, Koller JM, Snyder AZ, Campbell MC, Earhart GM, Perlmutter JS. Functional Connectivity of Vermis Correlates with Future Gait Impairments in Parkinson's Disease. Mov Disord. 2021 Nov;36(11):2559-2568. doi: 10.1002/mds.28684. Epub 2021 Jun 10. PMID 34109682
- [Background] Nemanich ST, McNeely ME, Earhart GM, Norris SA, Black KJ. A Case of Apparent Upper-Body Freezing in Parkinsonism while Using a Wheelchair. Front Neurol. 2017 May 15;8:205. doi: 10.3389/fneur.2017.00205. eCollection 2017. PMID 28555128
- [Background] Horin AP, Harrison EC, Rawson KS, Earhart GM. People with Parkinson disease with and without freezing of gait respond similarly to external and self-generated cues. Gait Posture. 2020 Oct;82:161-166. doi: 10.1016/j.gaitpost.2020.09.005. Epub 2020 Sep 6. PMID 32932076
- [Background] Baudendistel ST, Haussler AM, Rawson KS, Earhart GM. Minimal clinically important differences of spatiotemporal gait variables in Parkinson disease. Gait Posture. 2024 Feb;108:257-263. doi: 10.1016/j.gaitpost.2023.11.016. Epub 2023 Nov 25. PMID 38150946
- [Background] Girnis JL, Cavanaugh JT, Baker TC, Duncan RP, Fulford D, LaValley MP, Lawrence M, Nordahl T, Porciuncula F, Rawson KS, Saint-Hilaire M, Thomas CA, Zajac JA, Earhart GM, Ellis TD. Natural Walking Intensity in Persons With Parkinson Disease. J Neurol Phys Ther. 2023 Jul 1;47(3):146-154. doi: 10.1097/NPT.0000000000000440. Epub 2023 Apr 4. PMID 37016469
- [Background] Zajac JA, Cavanaugh JT, Baker T, Duncan RP, Fulford D, Girnis J, LaValley M, Nordahl T, Porciuncula F, Rawson KS, Saint-Hilaire M, Thomas CA, Earhart GM, Ellis TD. Does clinically measured walking capacity contribute to real-world walking performance in Parkinson's disease? Parkinsonism Relat Disord. 2022 Dec;105:123-127. doi: 10.1016/j.parkreldis.2022.11.016. Epub 2022 Nov 15. PMID 36423521
- [Background] Rawson KS, McNeely ME, Duncan RP, Pickett KA, Perlmutter JS, Earhart GM. Exercise and Parkinson Disease: Comparing Tango, Treadmill, and Stretching. J Neurol Phys Ther. 2019 Jan;43(1):26-32. doi: 10.1097/NPT.0000000000000245. PMID 30531383
- [Background] Younce JR, Campbell MC, Perlmutter JS, Norris SA. Thalamic and ventricular volumes predict motor response to deep brain stimulation for Parkinson's disease. Parkinsonism Relat Disord. 2019 Apr;61:64-69. doi: 10.1016/j.parkreldis.2018.11.026. Epub 2018 Nov 28. PMID 30527905
- [Background] Gordon EM, May GJ, Nelson SM. MRI-based measures of intracortical myelin are sensitive to a history of TBI and are associated with functional connectivity. Neuroimage. 2019 Oct 15;200:199-209. doi: 10.1016/j.neuroimage.2019.06.026. Epub 2019 Jun 13. PMID 31203023
- [Background] Rajesh A, Seider NA, Newbold DJ, Adeyemo B, Marek S, Greene DJ, Snyder AZ, Shimony JS, Laumann TO, Dosenbach NUF, Gordon EM. Structure-function coupling in highly sampled individual brains. Cereb Cortex. 2024 Sep 3;34(9):bhae361. doi: 10.1093/cercor/bhae361. PMID 39277800
- [Background] Zheng A, Montez DF, Marek S, Gilmore AW, Newbold DJ, Laumann TO, Kay BP, Seider NA, Van AN, Hampton JM, Alexopoulos D, Schlaggar BL, Sylvester CM, Greene DJ, Shimony JS, Nelson SM, Wig GS, Gratton C, McDermott KB, Raichle ME, Gordon EM, Dosenbach NUF. Parallel hippocampal-parietal circuits for self- and goal-oriented processing. Proc Natl Acad Sci U S A. 2021 Aug 24;118(34):e2101743118. doi: 10.1073/pnas.2101743118. PMID 34404728
- [Background] Gordon EM, Laumann TO, Marek S, Raut RV, Gratton C, Newbold DJ, Greene DJ, Coalson RS, Snyder AZ, Schlaggar BL, Petersen SE, Dosenbach NUF, Nelson SM. Default-mode network streams for coupling to language and control systems. Proc Natl Acad Sci U S A. 2020 Jul 21;117(29):17308-17319. doi: 10.1073/pnas.2005238117. Epub 2020 Jul 6. PMID 32632019
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Campbell MC, Myers PS, Weigand AJ, Foster ER, Cairns NJ, Jackson JJ, Lessov-Schlaggar CN, Perlmutter JS. Parkinson disease clinical subtypes: key features & clinical milestones. Ann Clin Transl Neurol. 2020 Aug;7(8):1272-1283. doi: 10.1002/acn3.51102. Epub 2020 Jun 29. PMID 32602253
- [Background] Myers PS, Jackson JJ, Clover AK, Lessov-Schlaggar CN, Foster ER, Maiti B, Perlmutter JS, Campbell MC. Distinct progression patterns across Parkinson disease clinical subtypes. Ann Clin Transl Neurol. 2021 Aug;8(8):1695-1708. doi: 10.1002/acn3.51436. Epub 2021 Jul 26. PMID 34310084
- [Background] Ciric R, Wolf DH, Power JD, Roalf DR, Baum GL, Ruparel K, Shinohara RT, Elliott MA, Eickhoff SB, Davatzikos C, Gur RC, Gur RE, Bassett DS, Satterthwaite TD. Benchmarking of participant-level confound regression strategies for the control of motion artifact in studies of functional connectivity. Neuroimage. 2017 Jul 1;154:174-187. doi: 10.1016/j.neuroimage.2017.03.020. Epub 2017 Mar 14. PMID 28302591
- [Background] Fan YS, Li L, Peng Y, Li H, Guo J, Li M, Yang S, Yao M, Zhao J, Liu H, Liao W, Guo X, Han S, Cui Q, Duan X, Xu Y, Zhang Y, Chen H. Individual-specific functional connectome biomarkers predict schizophrenia positive symptoms during adolescent brain maturation. Hum Brain Mapp. 2020 Dec 2;42(5):1475-84. doi: 10.1002/hbm.25307. Online ahead of print. PMID 33289223
- [Background] Brennan BP, Wang D, Li M, Perriello C, Ren J, Elias JA, Van Kirk NP, Krompinger JW, Pope HG Jr, Haber SN, Rauch SL, Baker JT, Liu H. Use of an Individual-Level Approach to Identify Cortical Connectivity Biomarkers in Obsessive-Compulsive Disorder. Biol Psychiatry Cogn Neurosci Neuroimaging. 2019 Jan;4(1):27-38. doi: 10.1016/j.bpsc.2018.07.014. Epub 2018 Aug 16. PMID 30262337
- [Background] Lynch CJ, Elbau I, Ng T, Ayaz A, Zhu S, Manfredi N, Johnson M, Wolk D, Power JD, Gordon EM, Kay K, Aloysi A, Moia S, Caballero-Gaudes C, Victoria LW, Solomonov N, Goldwaser E, Zebley B, Grosenick L, Downar J, Vila-Rodriguez F, Daskalakis ZJ, Blumberger DM, Williams N, Gunning FM, Liston C. Expansion of a frontostriatal salience network in individuals with depression. bioRxiv [Preprint]. 2023 Aug 14:2023.08.09.551651. doi: 10.1101/2023.08.09.551651. PMID 37645792
- [Background] Seider NA, Adeyemo B, Miller R, Newbold DJ, Hampton JM, Scheidter KM, Rutlin J, Laumann TO, Roland JL, Montez DF, Van AN, Zheng A, Marek S, Kay BP, Bretthorst GL, Schlaggar BL, Greene DJ, Wang Y, Petersen SE, Barch DM, Gordon EM, Snyder AZ, Shimony JS, Dosenbach NUF. Accuracy and reliability of diffusion imaging models. Neuroimage. 2022 Jul 1;254:119138. doi: 10.1016/j.neuroimage.2022.119138. Epub 2022 Mar 23. PMID 35339687
- [Background] Horn A, Reich M, Vorwerk J, Li N, Wenzel G, Fang Q, Schmitz-Hubsch T, Nickl R, Kupsch A, Volkmann J, Kuhn AA, Fox MD. Connectivity Predicts deep brain stimulation outcome in Parkinson disease. Ann Neurol. 2017 Jul;82(1):67-78. doi: 10.1002/ana.24974. PMID 28586141
- [Background] Coenen VA, Madler B, Schiffbauer H, Urbach H, Allert N. Individual fiber anatomy of the subthalamic region revealed with diffusion tensor imaging: a concept to identify the deep brain stimulation target for tremor suppression. Neurosurgery. 2011 Apr;68(4):1069-75; discussion 1075-6. doi: 10.1227/NEU.0b013e31820a1a20. PMID 21242831
- [Background] Horn A, Li N, Dembek TA, Kappel A, Boulay C, Ewert S, Tietze A, Husch A, Perera T, Neumann WJ, Reisert M, Si H, Oostenveld R, Rorden C, Yeh FC, Fang Q, Herrington TM, Vorwerk J, Kuhn AA. Lead-DBS v2: Towards a comprehensive pipeline for deep brain stimulation imaging. Neuroimage. 2019 Jan 1;184:293-316. doi: 10.1016/j.neuroimage.2018.08.068. Epub 2018 Sep 1. PMID 30179717
- [Background] Stevens AK, Blanchard BE, Talley AE, Brown JL, Halvorson MA, Janssen T, King KM, Littlefield AK. State-Level Impulsivity, Affect, and Alcohol: A Psychometric Evaluation of the Momentary Impulsivity Scale Across Two Intensive Longitudinal Samples. J Res Pers. 2020 Apr;85:103914. doi: 10.1016/j.jrp.2020.103914. Epub 2020 Jan 15. PMID 32341603
- [Background] Johnson PC, Barry SJ, Ferguson HM, Muller P. Power analysis for generalized linear mixed models in ecology and evolution. Methods Ecol Evol. 2015 Feb;6(2):133-142. doi: 10.1111/2041-210X.12306. Epub 2014 Dec 6. PMID 25893088
- [Background] Ren J, Ren W, Zhou Y, Dahmani L, Duan X, Fu X, Wang Y, Pan R, Zhao J, Zhang P, Wang B, Yu W, Chen Z, Zhang X, Sun J, Ding M, Huang J, Xu L, Li S, Wang W, Xie W, Zhang H, Liu H. Personalized functional imaging-guided rTMS on the superior frontal gyrus for post-stroke aphasia: A randomized sham-controlled trial. Brain Stimul. 2023 Sep-Oct;16(5):1313-1321. doi: 10.1016/j.brs.2023.08.023. Epub 2023 Aug 29. PMID 37652135
- [Background] Prateek GV, Mazzoni P, Earhart GM, Nehorai A. Gait Cycle Validation and Segmentation Using Inertial Sensors. IEEE Trans Biomed Eng. 2020 Aug;67(8):2132-2144. doi: 10.1109/TBME.2019.2955423. Epub 2019 Nov 25. PMID 31765301
- [Background] Prateek GV, Skog I, McNeely ME, Duncan RP, Earhart GM, Nehorai A. Modeling, Detecting, and Tracking Freezing of Gait in Parkinson Disease Using Inertial Sensors. IEEE Trans Biomed Eng. 2018 Oct;65(10):2152-2161. doi: 10.1109/TBME.2017.2785625. Epub 2017 Dec 20. PMID 29989948
- [Background] Rosvall M, Bergstrom CT. Maps of random walks on complex networks reveal community structure. Proc Natl Acad Sci U S A. 2008 Jan 29;105(4):1118-23. doi: 10.1073/pnas.0706851105. Epub 2008 Jan 23. PMID 18216267
- [Background] Gratton C, Dworetsky A, Coalson RS, Adeyemo B, Laumann TO, Wig GS, Kong TS, Gratton G, Fabiani M, Barch DM, Tranel D, Miranda-Dominguez O, Fair DA, Dosenbach NUF, Snyder AZ, Perlmutter JS, Petersen SE, Campbell MC. Removal of high frequency contamination from motion estimates in single-band fMRI saves data without biasing functional connectivity. Neuroimage. 2020 Aug 15;217:116866. doi: 10.1016/j.neuroimage.2020.116866. Epub 2020 Apr 20. PMID 32325210
- [Background] Siegel JS, Mitra A, Laumann TO, Seitzman BA, Raichle M, Corbetta M, Snyder AZ. Data Quality Influences Observed Links Between Functional Connectivity and Behavior. Cereb Cortex. 2017 Sep 1;27(9):4492-4502. doi: 10.1093/cercor/bhw253. PMID 27550863
- [Background] Power JD, Mitra A, Laumann TO, Snyder AZ, Schlaggar BL, Petersen SE. Methods to detect, characterize, and remove motion artifact in resting state fMRI. Neuroimage. 2014 Jan 1;84:320-41. doi: 10.1016/j.neuroimage.2013.08.048. Epub 2013 Aug 29. PMID 23994314
- [Background] Power JD, Barnes KA, Snyder AZ, Schlaggar BL, Petersen SE. Spurious but systematic correlations in functional connectivity MRI networks arise from subject motion. Neuroimage. 2012 Feb 1;59(3):2142-54. doi: 10.1016/j.neuroimage.2011.10.018. Epub 2011 Oct 14. PMID 22019881
- [Background] Marcus DS, Harwell J, Olsen T, Hodge M, Glasser MF, Prior F, Jenkinson M, Laumann T, Curtiss SW, Van Essen DC. Informatics and data mining tools and strategies for the human connectome project. Front Neuroinform. 2011 Jun 27;5:4. doi: 10.3389/fninf.2011.00004. eCollection 2011. PMID 21743807
- [Background] Newbold DJ, Laumann TO, Hoyt CR, Hampton JM, Montez DF, Raut RV, Ortega M, Mitra A, Nielsen AN, Miller DB, Adeyemo B, Nguyen AL, Scheidter KM, Tanenbaum AB, Van AN, Marek S, Schlaggar BL, Carter AR, Greene DJ, Gordon EM, Raichle ME, Petersen SE, Snyder AZ, Dosenbach NUF. Plasticity and Spontaneous Activity Pulses in Disused Human Brain Circuits. Neuron. 2020 Aug 5;107(3):580-589.e6. doi: 10.1016/j.neuron.2020.05.007. Epub 2020 Jun 16. PMID 32778224
- [Background] Greene DJ, Koller JM, Hampton JM, Wesevich V, Van AN, Nguyen AL, Hoyt CR, McIntyre L, Earl EA, Klein RL, Shimony JS, Petersen SE, Schlaggar BL, Fair DA, Dosenbach NUF. Behavioral interventions for reducing head motion during MRI scans in children. Neuroimage. 2018 May 1;171:234-245. doi: 10.1016/j.neuroimage.2018.01.023. Epub 2018 Jan 12. PMID 29337280
- [Background] Dosenbach NUF, Koller JM, Earl EA, Miranda-Dominguez O, Klein RL, Van AN, Snyder AZ, Nagel BJ, Nigg JT, Nguyen AL, Wesevich V, Greene DJ, Fair DA. Real-time motion analytics during brain MRI improve data quality and reduce costs. Neuroimage. 2017 Nov 1;161:80-93. doi: 10.1016/j.neuroimage.2017.08.025. Epub 2017 Aug 10. PMID 28803940
- [Background] Weintraub D, Hoops S, Shea JA, Lyons KE, Pahwa R, Driver-Dunckley ED, Adler CH, Potenza MN, Miyasaki J, Siderowf AD, Duda JE, Hurtig HI, Colcher A, Horn SS, Stern MB, Voon V. Validation of the questionnaire for impulsive-compulsive disorders in Parkinson's disease. Mov Disord. 2009 Jul 30;24(10):1461-7. doi: 10.1002/mds.22571. PMID 19452562
- [Background] Shine JM, Mills JMZ, Qiu J, O'Callaghan C, Terpening Z, Halliday GM, Naismith SL, Lewis SJG. Validation of the Psychosis and Hallucinations Questionnaire in Non-demented Patients with Parkinson's Disease. Mov Disord Clin Pract. 2015 Mar 16;2(2):175-181. doi: 10.1002/mdc3.12139. eCollection 2015 Jun. PMID 30363832
- [Background] Grace J, Stout JC, Malloy PF. Assessing frontal lobe behavioral syndromes with the frontal lobe personality scale. Assessment. 1999 Sep;6(3):269-84. doi: 10.1177/107319119900600307. PMID 10445964
- [Background] Marin RS, Biedrzycki RC, Firinciogullari S. Reliability and validity of the Apathy Evaluation Scale. Psychiatry Res. 1991 Aug;38(2):143-62. doi: 10.1016/0165-1781(91)90040-v. PMID 1754629
- [Background] Spielberger CD, Vagg PR. Psychometric properties of the STAI: a reply to Ramanaiah, Franzen, and Schill. J Pers Assess. 1984 Feb;48(1):95-7. doi: 10.1207/s15327752jpa4801_16. No abstract available. PMID 6707862
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Cohen RG, Klein KA, Nomura M, Fleming M, Mancini M, Giladi N, Nutt JG, Horak FB. Inhibition, executive function, and freezing of gait. J Parkinsons Dis. 2014;4(1):111-22. doi: 10.3233/JPD-130221. PMID 24496099
- [Background] Obeso I, Wilkinson L, Casabona E, Speekenbrink M, Luisa Bringas M, Alvarez M, Alvarez L, Pavon N, Rodriguez-Oroz MC, Macias R, Obeso JA, Jahanshahi M. The subthalamic nucleus and inhibitory control: impact of subthalamotomy in Parkinson's disease. Brain. 2014 May;137(Pt 5):1470-80. doi: 10.1093/brain/awu058. Epub 2014 Mar 22. PMID 24657985
- [Background] Obeso I, Wilkinson L, Casabona E, Bringas ML, Alvarez M, Alvarez L, Pavon N, Rodriguez-Oroz MC, Macias R, Obeso JA, Jahanshahi M. Deficits in inhibitory control and conflict resolution on cognitive and motor tasks in Parkinson's disease. Exp Brain Res. 2011 Jul;212(3):371-84. doi: 10.1007/s00221-011-2736-6. Epub 2011 Jun 4. PMID 21643718
- [Background] Donders FC. On the speed of mental processes. Acta Psychol (Amst). 1969;30:412-31. doi: 10.1016/0001-6918(69)90065-1. No abstract available. PMID 5811531
- [Background] Aron AR, Behrens TE, Smith S, Frank MJ, Poldrack RA. Triangulating a cognitive control network using diffusion-weighted magnetic resonance imaging (MRI) and functional MRI. J Neurosci. 2007 Apr 4;27(14):3743-52. doi: 10.1523/JNEUROSCI.0519-07.2007. PMID 17409238
- [Background] May DS, Tueth LE, Earhart GM, Mazzoni P. Using Wearable Sensors to Assess Freezing of Gait in the Real World. Bioengineering (Basel). 2023 Feb 23;10(3):289. doi: 10.3390/bioengineering10030289. PMID 36978680
- [Background] Webster KE, Wittwer JE, Feller JA. Validity of the GAITRite walkway system for the measurement of averaged and individual step parameters of gait. Gait Posture. 2005 Dec;22(4):317-21. doi: 10.1016/j.gaitpost.2004.10.005. Epub 2004 Dec 10. PMID 16274913
- [Background] Bilney B, Morris M, Webster K. Concurrent related validity of the GAITRite walkway system for quantification of the spatial and temporal parameters of gait. Gait Posture. 2003 Feb;17(1):68-74. doi: 10.1016/s0966-6362(02)00053-x. PMID 12535728
- [Background] Tomlinson CL, Stowe R, Patel S, Rick C, Gray R, Clarke CE. Systematic review of levodopa dose equivalency reporting in Parkinson's disease. Mov Disord. 2010 Nov 15;25(15):2649-53. doi: 10.1002/mds.23429. PMID 21069833
- [Background] Nieuwboer A, Rochester L, Herman T, Vandenberghe W, Emil GE, Thomaes T, Giladi N. Reliability of the new freezing of gait questionnaire: agreement between patients with Parkinson's disease and their carers. Gait Posture. 2009 Nov;30(4):459-63. doi: 10.1016/j.gaitpost.2009.07.108. Epub 2009 Aug 5. PMID 19660949
- [Background] Gill DJ, Freshman A, Blender JA, Ravina B. The Montreal cognitive assessment as a screening tool for cognitive impairment in Parkinson's disease. Mov Disord. 2008 May 15;23(7):1043-1046. doi: 10.1002/mds.22017. PMID 18381646
- [Background] Emre M, Aarsland D, Brown R, Burn DJ, Duyckaerts C, Mizuno Y, Broe GA, Cummings J, Dickson DW, Gauthier S, Goldman J, Goetz C, Korczyn A, Lees A, Levy R, Litvan I, McKeith I, Olanow W, Poewe W, Quinn N, Sampaio C, Tolosa E, Dubois B. Clinical diagnostic criteria for dementia associated with Parkinson's disease. Mov Disord. 2007 Sep 15;22(12):1689-707; quiz 1837. doi: 10.1002/mds.21507. PMID 17542011
- [Background] Racette BA, Rundle M, Parsian A, Perlmutter JS. Evaluation of a screening questionnaire for genetic studies of Parkinson's disease. Am J Med Genet. 1999 Oct 15;88(5):539-43. PMID 10490713
- [Background] Younce JR, Campbell MC, Hershey T, Tanenbaum AB, Milchenko M, Ushe M, Karimi M, Tabbal SD, Kim AE, Snyder AZ, Perlmutter JS, Norris SA. Resting-State Functional Connectivity Predicts STN DBS Clinical Response. Mov Disord. 2021 Mar;36(3):662-671. doi: 10.1002/mds.28376. Epub 2020 Nov 19. PMID 33211330
- [Background] Maiti B, Koller JM, Snyder AZ, Tanenbaum AB, Norris SA, Campbell MC, Perlmutter JS. Cognitive correlates of cerebellar resting-state functional connectivity in Parkinson disease. Neurology. 2020 Jan 28;94(4):e384-e396. doi: 10.1212/WNL.0000000000008754. Epub 2019 Dec 17. PMID 31848257
- [Background] Gordon EM, Scheibel RS, Zambrano-Vazquez L, Jia-Richards M, May GJ, Meyer EC, Nelson SM. High-Fidelity Measures of Whole-Brain Functional Connectivity and White Matter Integrity Mediate Relationships between Traumatic Brain Injury and Post-Traumatic Stress Disorder Symptoms. J Neurotrauma. 2018 Mar 1;35(5):767-779. doi: 10.1089/neu.2017.5428. Epub 2018 Jan 29. PMID 29179667
- [Background] Seitzman BA, Gratton C, Laumann TO, Gordon EM, Adeyemo B, Dworetsky A, Kraus BT, Gilmore AW, Berg JJ, Ortega M, Nguyen A, Greene DJ, McDermott KB, Nelson SM, Lessov-Schlaggar CN, Schlaggar BL, Dosenbach NUF, Petersen SE. Trait-like variants in human functional brain networks. Proc Natl Acad Sci U S A. 2019 Nov 5;116(45):22851-22861. doi: 10.1073/pnas.1902932116. Epub 2019 Oct 14. PMID 31611415
- [Background] Gratton C, Laumann TO, Nielsen AN, Greene DJ, Gordon EM, Gilmore AW, Nelson SM, Coalson RS, Snyder AZ, Schlaggar BL, Dosenbach NUF, Petersen SE. Functional Brain Networks Are Dominated by Stable Group and Individual Factors, Not Cognitive or Daily Variation. Neuron. 2018 Apr 18;98(2):439-452.e5. doi: 10.1016/j.neuron.2018.03.035. PMID 29673485
- [Background] Bianciardi M, Toschi N, Edlow BL, Eichner C, Setsompop K, Polimeni JR, Brown EN, Kinney HC, Rosen BR, Wald LL. Toward an In Vivo Neuroimaging Template of Human Brainstem Nuclei of the Ascending Arousal, Autonomic, and Motor Systems. Brain Connect. 2015 Dec;5(10):597-607. doi: 10.1089/brain.2015.0347. Epub 2015 Aug 11. PMID 26066023
- [Background] Van AN, Montez DF, Laumann TO, Suljic V, Madison T, Baden NJ, Ramirez-Perez N, Scheidter KM, Monk JS, Whiting FI, Adeyemo B, Chauvin RJ, Krimmel SR, Metoki A, Rajesh A, Roland JL, Salo T, Wang A, Weldon KB, Sotiras A, Shimony JS, Kay BP, Nelson SM, Tervo-Clemmens B, Marek SA, Vizioli L, Yacoub E, Satterthwaite TD, Gordon EM, Fair DA, Tisdall MD, Dosenbach NUF. Framewise multi-echo distortion correction for superior functional MRI. bioRxiv [Preprint]. 2023 Nov 29:2023.11.28.568744. doi: 10.1101/2023.11.28.568744. PMID 38077010
- [Background] Dowdle LT, Vizioli L, Moeller S, Akcakaya M, Olman C, Ghose G, Yacoub E, Ugurbil K. Evaluating increases in sensitivity from NORDIC for diverse fMRI acquisition strategies. Neuroimage. 2023 Apr 15;270:119949. doi: 10.1016/j.neuroimage.2023.119949. Epub 2023 Feb 17. PMID 36804422
- [Background] Vizioli L, Moeller S, Dowdle L, Akcakaya M, De Martino F, Yacoub E, Ugurbil K. Lowering the thermal noise barrier in functional brain mapping with magnetic resonance imaging. Nat Commun. 2021 Aug 30;12(1):5181. doi: 10.1038/s41467-021-25431-8. PMID 34462435
- [Background] Lynch CJ, Power JD, Scult MA, Dubin M, Gunning FM, Liston C. Rapid Precision Functional Mapping of Individuals Using Multi-Echo fMRI. Cell Rep. 2020 Dec 22;33(12):108540. doi: 10.1016/j.celrep.2020.108540. PMID 33357444
- [Background] Kundu P, Brenowitz ND, Voon V, Worbe Y, Vertes PE, Inati SJ, Saad ZS, Bandettini PA, Bullmore ET. Integrated strategy for improving functional connectivity mapping using multiecho fMRI. Proc Natl Acad Sci U S A. 2013 Oct 1;110(40):16187-92. doi: 10.1073/pnas.1301725110. Epub 2013 Sep 13. PMID 24038744
- [Background] Kundu P, Inati SJ, Evans JW, Luh WM, Bandettini PA. Differentiating BOLD and non-BOLD signals in fMRI time series using multi-echo EPI. Neuroimage. 2012 Apr 15;60(3):1759-70. doi: 10.1016/j.neuroimage.2011.12.028. Epub 2011 Dec 23. PMID 22209809
- [Background] Haynes WI, Haber SN. The organization of prefrontal-subthalamic inputs in primates provides an anatomical substrate for both functional specificity and integration: implications for Basal Ganglia models and deep brain stimulation. J Neurosci. 2013 Mar 13;33(11):4804-14. doi: 10.1523/JNEUROSCI.4674-12.2013. PMID 23486951
- [Background] Haber SN, Calzavara R. The cortico-basal ganglia integrative network: the role of the thalamus. Brain Res Bull. 2009 Feb 16;78(2-3):69-74. doi: 10.1016/j.brainresbull.2008.09.013. Epub 2008 Oct 23. PMID 18950692
- [Background] Haber SN. The primate basal ganglia: parallel and integrative networks. J Chem Neuroanat. 2003 Dec;26(4):317-30. doi: 10.1016/j.jchemneu.2003.10.003. PMID 14729134
- [Background] Haber SN. Corticostriatal circuitry. Dialogues Clin Neurosci. 2016 Mar;18(1):7-21. doi: 10.31887/DCNS.2016.18.1/shaber. PMID 27069376
- [Background] Noble S, Spann MN, Tokoglu F, Shen X, Constable RT, Scheinost D. Influences on the Test-Retest Reliability of Functional Connectivity MRI and its Relationship with Behavioral Utility. Cereb Cortex. 2017 Nov 1;27(11):5415-5429. doi: 10.1093/cercor/bhx230. PMID 28968754
- [Background] Krimmel SR, Laumann TO, Chauvin RJ, Hershey T, Roland JL, Shimony JS, Willie JT, Norris SA, Marek S, Van AN, Monk J, Scheidter KM, Whiting F, Ramirez-Perez N, Metoki A, Wang A, Kay BP, Nahman-Averbuch H, Fair DA, Lynch CJ, Raichle ME, Gordon EM, Dosenbach NUF. The brainstem's red nucleus was evolutionarily upgraded to support goal-directed action. bioRxiv [Preprint]. 2024 Jan 1:2023.12.30.573730. doi: 10.1101/2023.12.30.573730. PMID 38260662
- [Background] Gordon EM, Laumann TO, Marek S, Newbold DJ, Hampton JM, Seider NA, Montez DF, Nielsen AM, Van AN, Zheng A, Miller R, Siegel JS, Kay BP, Snyder AZ, Greene DJ, Schlaggar BL, Petersen SE, Nelson SM, Dosenbach NUF. Individualized Functional Subnetworks Connect Human Striatum and Frontal Cortex. Cereb Cortex. 2022 Jun 16;32(13):2868-2884. doi: 10.1093/cercor/bhab387. PMID 34718460
- [Background] Laumann TO, Zorumski CF, Dosenbach NUF. Precision Neuroimaging for Localization-Related Psychiatry. JAMA Psychiatry. 2023 Aug 1;80(8):763-764. doi: 10.1001/jamapsychiatry.2023.1576. PMID 37285163
- [Background] Gratton C, Kraus BT, Greene DJ, Gordon EM, Laumann TO, Nelson SM, Dosenbach NUF, Petersen SE. Defining Individual-Specific Functional Neuroanatomy for Precision Psychiatry. Biol Psychiatry. 2020 Jul 1;88(1):28-39. doi: 10.1016/j.biopsych.2019.10.026. Epub 2019 Nov 7. PMID 31916942
- [Background] Gordon EM, Lynch CJ, Gratton C, Laumann TO, Gilmore AW, Greene DJ, Ortega M, Nguyen AL, Schlaggar BL, Petersen SE, Dosenbach NUF, Nelson SM. Three Distinct Sets of Connector Hubs Integrate Human Brain Function. Cell Rep. 2018 Aug 14;24(7):1687-1695.e4. doi: 10.1016/j.celrep.2018.07.050. PMID 30110625
- [Background] Bijsterbosch JD, Woolrich MW, Glasser MF, Robinson EC, Beckmann CF, Van Essen DC, Harrison SJ, Smith SM. The relationship between spatial configuration and functional connectivity of brain regions. Elife. 2018 Feb 16;7:e32992. doi: 10.7554/eLife.32992. PMID 29451491
- [Background] Laumann TO, Gordon EM, Adeyemo B, Snyder AZ, Joo SJ, Chen MY, Gilmore AW, McDermott KB, Nelson SM, Dosenbach NU, Schlaggar BL, Mumford JA, Poldrack RA, Petersen SE. Functional System and Areal Organization of a Highly Sampled Individual Human Brain. Neuron. 2015 Aug 5;87(3):657-70. doi: 10.1016/j.neuron.2015.06.037. Epub 2015 Jul 23. PMID 26212711
- [Background] Wang D, Buckner RL, Fox MD, Holt DJ, Holmes AJ, Stoecklein S, Langs G, Pan R, Qian T, Li K, Baker JT, Stufflebeam SM, Wang K, Wang X, Hong B, Liu H. Parcellating cortical functional networks in individuals. Nat Neurosci. 2015 Dec;18(12):1853-60. doi: 10.1038/nn.4164. Epub 2015 Nov 9. PMID 26551545
- [Background] Braga RM, Buckner RL. Parallel Interdigitated Distributed Networks within the Individual Estimated by Intrinsic Functional Connectivity. Neuron. 2017 Jul 19;95(2):457-471.e5. doi: 10.1016/j.neuron.2017.06.038. PMID 28728026
- [Background] Gordon EM, Laumann TO, Adeyemo B, Gilmore AW, Nelson SM, Dosenbach NUF, Petersen SE. Individual-specific features of brain systems identified with resting state functional correlations. Neuroimage. 2017 Feb 1;146:918-939. doi: 10.1016/j.neuroimage.2016.08.032. Epub 2016 Sep 15. PMID 27640749
- [Background] Gordon EM, Laumann TO, Adeyemo B, Petersen SE. Individual Variability of the System-Level Organization of the Human Brain. Cereb Cortex. 2017 Jan 1;27(1):386-399. doi: 10.1093/cercor/bhv239. PMID 26464473
- [Background] Manza P, Zhang S, Li CS, Leung HC. Resting-state functional connectivity of the striatum in early-stage Parkinson's disease: Cognitive decline and motor symptomatology. Hum Brain Mapp. 2016 Feb;37(2):648-62. doi: 10.1002/hbm.23056. Epub 2015 Nov 14. PMID 26566885
- [Background] Baggio HC, Segura B, Garrido-Millan JL, Marti MJ, Compta Y, Valldeoriola F, Tolosa E, Junque C. Resting-state frontostriatal functional connectivity in Parkinson's disease-related apathy. Mov Disord. 2015 Apr 15;30(5):671-9. doi: 10.1002/mds.26137. Epub 2015 Jan 20. PMID 25600482
- [Background] Kwak Y, Peltier S, Bohnen NI, Muller ML, Dayalu P, Seidler RD. Altered resting state cortico-striatal connectivity in mild to moderate stage Parkinson's disease. Front Syst Neurosci. 2010 Sep 15;4:143. doi: 10.3389/fnsys.2010.00143. eCollection 2010. PMID 21206528
- [Background] Helmich RC, Derikx LC, Bakker M, Scheeringa R, Bloem BR, Toni I. Spatial remapping of cortico-striatal connectivity in Parkinson's disease. Cereb Cortex. 2010 May;20(5):1175-86. doi: 10.1093/cercor/bhp178. Epub 2009 Aug 26. PMID 19710357
- [Background] Wu T, Long X, Wang L, Hallett M, Zang Y, Li K, Chan P. Functional connectivity of cortical motor areas in the resting state in Parkinson's disease. Hum Brain Mapp. 2011 Sep;32(9):1443-57. doi: 10.1002/hbm.21118. Epub 2010 Aug 25. PMID 20740649
- [Background] Wu T, Wang L, Chen Y, Zhao C, Li K, Chan P. Changes of functional connectivity of the motor network in the resting state in Parkinson's disease. Neurosci Lett. 2009 Aug 21;460(1):6-10. doi: 10.1016/j.neulet.2009.05.046. Epub 2009 May 20. PMID 19463891
- [Background] Hacker CD, Perlmutter JS, Criswell SR, Ances BM, Snyder AZ. Resting state functional connectivity of the striatum in Parkinson's disease. Brain. 2012 Dec;135(Pt 12):3699-711. doi: 10.1093/brain/aws281. Epub 2012 Nov 28. PMID 23195207
- [Background] de Schipper LJ, Hafkemeijer A, van der Grond J, Marinus J, Henselmans JML, van Hilten JJ. Altered Whole-Brain and Network-Based Functional Connectivity in Parkinson's Disease. Front Neurol. 2018 Jun 6;9:419. doi: 10.3389/fneur.2018.00419. eCollection 2018. PMID 29928255
- [Background] Tessitore A, Cirillo M, De Micco R. Functional Connectivity Signatures of Parkinson's Disease. J Parkinsons Dis. 2019;9(4):637-652. doi: 10.3233/JPD-191592. PMID 31450512
- [Background] Gratton C, Koller JM, Shannon W, Greene DJ, Maiti B, Snyder AZ, Petersen SE, Perlmutter JS, Campbell MC. Emergent Functional Network Effects in Parkinson Disease. Cereb Cortex. 2019 Apr 1;29(4):1701. doi: 10.1093/cercor/bhy229. No abstract available. PMID 30418543
- [Background] Fox MD, Greicius M. Clinical applications of resting state functional connectivity. Front Syst Neurosci. 2010 Jun 17;4:19. doi: 10.3389/fnsys.2010.00019. eCollection 2010. PMID 20592951
- [Background] Greene DJ, Marek S, Gordon EM, Siegel JS, Gratton C, Laumann TO, Gilmore AW, Berg JJ, Nguyen AL, Dierker D, Van AN, Ortega M, Newbold DJ, Hampton JM, Nielsen AN, McDermott KB, Roland JL, Norris SA, Nelson SM, Snyder AZ, Schlaggar BL, Petersen SE, Dosenbach NUF. Integrative and Network-Specific Connectivity of the Basal Ganglia and Thalamus Defined in Individuals. Neuron. 2020 Feb 19;105(4):742-758.e6. doi: 10.1016/j.neuron.2019.11.012. Epub 2019 Dec 10. PMID 31836321
- [Background] Marek S, Siegel JS, Gordon EM, Raut RV, Gratton C, Newbold DJ, Ortega M, Laumann TO, Adeyemo B, Miller DB, Zheng A, Lopez KC, Berg JJ, Coalson RS, Nguyen AL, Dierker D, Van AN, Hoyt CR, McDermott KB, Norris SA, Shimony JS, Snyder AZ, Nelson SM, Barch DM, Schlaggar BL, Raichle ME, Petersen SE, Greene DJ, Dosenbach NUF. Spatial and Temporal Organization of the Individual Human Cerebellum. Neuron. 2018 Nov 21;100(4):977-993.e7. doi: 10.1016/j.neuron.2018.10.010. Epub 2018 Oct 25. PMID 30473014
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021
- [Background] Power JD, Cohen AL, Nelson SM, Wig GS, Barnes KA, Church JA, Vogel AC, Laumann TO, Miezin FM, Schlaggar BL, Petersen SE. Functional network organization of the human brain. Neuron. 2011 Nov 17;72(4):665-78. doi: 10.1016/j.neuron.2011.09.006. PMID 22099467
- [Background] Power JD, Schlaggar BL, Petersen SE. Studying brain organization via spontaneous fMRI signal. Neuron. 2014 Nov 19;84(4):681-96. doi: 10.1016/j.neuron.2014.09.007. Epub 2014 Nov 19. PMID 25459408
- [Background] Miranda-Dominguez O, Ragothaman A, Hermosillo R, Feczko E, Morris R, Carlson-Kuhta P, Nutt JG, Mancini M, Fair D, Horak FB. Lateralized Connectivity between Globus Pallidus and Motor Cortex is Associated with Freezing of Gait in Parkinson's Disease. Neuroscience. 2020 Sep 1;443:44-58. doi: 10.1016/j.neuroscience.2020.06.036. Epub 2020 Jul 3. PMID 32629155
- [Background] Fasano A, Laganiere SE, Lam S, Fox MD. Lesions causing freezing of gait localize to a cerebellar functional network. Ann Neurol. 2017 Jan;81(1):129-141. doi: 10.1002/ana.24845. PMID 28009063
- [Background] Levinthal DJ, Strick PL. Multiple areas of the cerebral cortex influence the stomach. Proc Natl Acad Sci U S A. 2020 Jun 9;117(23):13078-13083. doi: 10.1073/pnas.2002737117. Epub 2020 May 20. PMID 32434910
- [Background] Dum RP, Levinthal DJ, Strick PL. The mind-body problem: Circuits that link the cerebral cortex to the adrenal medulla. Proc Natl Acad Sci U S A. 2019 Dec 26;116(52):26321-26328. doi: 10.1073/pnas.1902297116. Epub 2019 Dec 23. PMID 31871146
- [Background] Dum RP, Levinthal DJ, Strick PL. Motor, cognitive, and affective areas of the cerebral cortex influence the adrenal medulla. Proc Natl Acad Sci U S A. 2016 Aug 30;113(35):9922-7. doi: 10.1073/pnas.1605044113. Epub 2016 Aug 15. PMID 27528671
- [Background] Paus T. Primate anterior cingulate cortex: where motor control, drive and cognition interface. Nat Rev Neurosci. 2001 Jun;2(6):417-24. doi: 10.1038/35077500. PMID 11389475
- [Background] Ebitz RB, Platt ML. Neuronal activity in primate dorsal anterior cingulate cortex signals task conflict and predicts adjustments in pupil-linked arousal. Neuron. 2015 Feb 4;85(3):628-40. doi: 10.1016/j.neuron.2014.12.053. PMID 25654259
- [Background] Critchley HD, Corfield DR, Chandler MP, Mathias CJ, Dolan RJ. Cerebral correlates of autonomic cardiovascular arousal: a functional neuroimaging investigation in humans. J Physiol. 2000 Feb 15;523 Pt 1(Pt 1):259-70. doi: 10.1111/j.1469-7793.2000.t01-1-00259.x. PMID 10673560
- [Background] Siegel JS, Snyder AZ, Metcalf NV, Fucetola RP, Hacker CD, Shimony JS, Shulman GL, Corbetta M. The circuitry of abulia: insights from functional connectivity MRI. Neuroimage Clin. 2014 Sep 23;6:320-6. doi: 10.1016/j.nicl.2014.09.012. eCollection 2014. PMID 25379445
- [Background] Srinivasan L, Asaad WF, Ginat DT, Gale JT, Dougherty DD, Williams ZM, Sejnowski TJ, Eskandar EN. Action initiation in the human dorsal anterior cingulate cortex. PLoS One. 2013;8(2):e55247. doi: 10.1371/journal.pone.0055247. Epub 2013 Feb 27. PMID 23460783
- [Background] Jensen MA, Huang H, Valencia GO, Klassen BT, van den Boom MA, Kaufmann TJ, Schalk G, Brunner P, Worrell GA, Hermes D, Miller KJ. A motor association area in the depths of the central sulcus. Nat Neurosci. 2023 Jul;26(7):1165-1169. doi: 10.1038/s41593-023-01346-z. Epub 2023 May 18. PMID 37202552
- [Background] Barch DM, Burgess GC, Harms MP, Petersen SE, Schlaggar BL, Corbetta M, Glasser MF, Curtiss S, Dixit S, Feldt C, Nolan D, Bryant E, Hartley T, Footer O, Bjork JM, Poldrack R, Smith S, Johansen-Berg H, Snyder AZ, Van Essen DC; WU-Minn HCP Consortium. Function in the human connectome: task-fMRI and individual differences in behavior. Neuroimage. 2013 Oct 15;80:169-89. doi: 10.1016/j.neuroimage.2013.05.033. Epub 2013 May 16. PMID 23684877
- [Background] Buckner RL, Krienen FM, Castellanos A, Diaz JC, Yeo BT. The organization of the human cerebellum estimated by intrinsic functional connectivity. J Neurophysiol. 2011 Nov;106(5):2322-45. doi: 10.1152/jn.00339.2011. Epub 2011 Jul 27. PMID 21795627
- [Background] Gordon EM, Laumann TO, Gilmore AW, Newbold DJ, Greene DJ, Berg JJ, Ortega M, Hoyt-Drazen C, Gratton C, Sun H, Hampton JM, Coalson RS, Nguyen AL, McDermott KB, Shimony JS, Snyder AZ, Schlaggar BL, Petersen SE, Nelson SM, Dosenbach NUF. Precision Functional Mapping of Individual Human Brains. Neuron. 2017 Aug 16;95(4):791-807.e7. doi: 10.1016/j.neuron.2017.07.011. Epub 2017 Jul 27. PMID 28757305
- [Background] Gordon EM, Chauvin RJ, Van AN, Rajesh A, Nielsen A, Newbold DJ, Lynch CJ, Seider NA, Krimmel SR, Scheidter KM, Monk J, Miller RL, Metoki A, Montez DF, Zheng A, Elbau I, Madison T, Nishino T, Myers MJ, Kaplan S, Badke D'Andrea C, Demeter DV, Feigelis M, Ramirez JSB, Xu T, Barch DM, Smyser CD, Rogers CE, Zimmermann J, Botteron KN, Pruett JR, Willie JT, Brunner P, Shimony JS, Kay BP, Marek S, Norris SA, Gratton C, Sylvester CM, Power JD, Liston C, Greene DJ, Roland JL, Petersen SE, Raichle ME, Laumann TO, Fair DA, Dosenbach NUF. A somato-cognitive action network alternates with effector regions in motor cortex. Nature. 2023 May;617(7960):351-359. doi: 10.1038/s41586-023-05964-2. Epub 2023 Apr 19. PMID 37076628
- [Background] Yu R, Liu B, Wang L, Chen J, Liu X. Enhanced functional connectivity between putamen and supplementary motor area in Parkinson's disease patients. PLoS One. 2013;8(3):e59717. doi: 10.1371/journal.pone.0059717. Epub 2013 Mar 26. PMID 23555758
- [Background] Playford ED, Jenkins IH, Passingham RE, Nutt J, Frackowiak RS, Brooks DJ. Impaired mesial frontal and putamen activation in Parkinson's disease: a positron emission tomography study. Ann Neurol. 1992 Aug;32(2):151-61. doi: 10.1002/ana.410320206. PMID 1510355
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Wang DD, de Hemptinne C, Miocinovic S, Ostrem JL, Galifianakis NB, San Luciano M, Starr PA. Pallidal Deep-Brain Stimulation Disrupts Pallidal Beta Oscillations and Coherence with Primary Motor Cortex in Parkinson's Disease. J Neurosci. 2018 May 9;38(19):4556-4568. doi: 10.1523/JNEUROSCI.0431-18.2018. Epub 2018 Apr 16. PMID 29661966
- [Background] Oswal A, Beudel M, Zrinzo L, Limousin P, Hariz M, Foltynie T, Litvak V, Brown P. Deep brain stimulation modulates synchrony within spatially and spectrally distinct resting state networks in Parkinson's disease. Brain. 2016 May;139(Pt 5):1482-96. doi: 10.1093/brain/aww048. Epub 2016 Mar 26. PMID 27017189
- [Background] Whitmer D, de Solages C, Hill B, Yu H, Henderson JM, Bronte-Stewart H. High frequency deep brain stimulation attenuates subthalamic and cortical rhythms in Parkinson's disease. Front Hum Neurosci. 2012 Jun 4;6:155. doi: 10.3389/fnhum.2012.00155. eCollection 2012. PMID 22675296
- [Background] Eusebio A, Thevathasan W, Doyle Gaynor L, Pogosyan A, Bye E, Foltynie T, Zrinzo L, Ashkan K, Aziz T, Brown P. Deep brain stimulation can suppress pathological synchronisation in parkinsonian patients. J Neurol Neurosurg Psychiatry. 2011 May;82(5):569-73. doi: 10.1136/jnnp.2010.217489. Epub 2010 Oct 9. PMID 20935326
- [Background] Shimamoto SA, Ryapolova-Webb ES, Ostrem JL, Galifianakis NB, Miller KJ, Starr PA. Subthalamic nucleus neurons are synchronized to primary motor cortex local field potentials in Parkinson's disease. J Neurosci. 2013 Apr 24;33(17):7220-33. doi: 10.1523/JNEUROSCI.4676-12.2013. PMID 23616531
- [Background] Lindenbach D, Bishop C. Critical involvement of the motor cortex in the pathophysiology and treatment of Parkinson's disease. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2737-50. doi: 10.1016/j.neubiorev.2013.09.008. Epub 2013 Oct 7. PMID 24113323
- [Background] Marreiros AC, Cagnan H, Moran RJ, Friston KJ, Brown P. Basal ganglia-cortical interactions in Parkinsonian patients. Neuroimage. 2013 Feb 1;66:301-10. doi: 10.1016/j.neuroimage.2012.10.088. Epub 2012 Nov 13. PMID 23153964
- [Background] Pavlides A, Hogan SJ, Bogacz R. Computational Models Describing Possible Mechanisms for Generation of Excessive Beta Oscillations in Parkinson's Disease. PLoS Comput Biol. 2015 Dec 18;11(12):e1004609. doi: 10.1371/journal.pcbi.1004609. eCollection 2015 Dec. PMID 26683341
- [Background] Oswal A, Cao C, Yeh CH, Neumann WJ, Gratwicke J, Akram H, Horn A, Li D, Zhan S, Zhang C, Wang Q, Zrinzo L, Foltynie T, Limousin P, Bogacz R, Sun B, Husain M, Brown P, Litvak V. Neural signatures of hyperdirect pathway activity in Parkinson's disease. Nat Commun. 2021 Aug 31;12(1):5185. doi: 10.1038/s41467-021-25366-0. PMID 34465771
- [Background] Kuhn AA, Kupsch A, Schneider GH, Brown P. Reduction in subthalamic 8-35 Hz oscillatory activity correlates with clinical improvement in Parkinson's disease. Eur J Neurosci. 2006 Apr;23(7):1956-60. doi: 10.1111/j.1460-9568.2006.04717.x. PMID 16623853
- [Background] Kuhn AA, Tsui A, Aziz T, Ray N, Brucke C, Kupsch A, Schneider GH, Brown P. Pathological synchronisation in the subthalamic nucleus of patients with Parkinson's disease relates to both bradykinesia and rigidity. Exp Neurol. 2009 Feb;215(2):380-7. doi: 10.1016/j.expneurol.2008.11.008. Epub 2008 Nov 25. PMID 19070616
- [Background] Brown P, Oliviero A, Mazzone P, Insola A, Tonali P, Di Lazzaro V. Dopamine dependency of oscillations between subthalamic nucleus and pallidum in Parkinson's disease. J Neurosci. 2001 Feb 1;21(3):1033-8. doi: 10.1523/JNEUROSCI.21-03-01033.2001. PMID 11157088
- [Background] Nonnekes J, Snijders AH, Nutt JG, Deuschl G, Giladi N, Bloem BR. Freezing of gait: a practical approach to management. Lancet Neurol. 2015 Jul;14(7):768-78. doi: 10.1016/S1474-4422(15)00041-1. Epub 2015 May 24. PMID 26018593
- [Background] Brozova H, Barnaure I, Ruzicka E, Stochl J, Alterman R, Tagliati M. Short- and Long-Term Effects of DBS on Gait in Parkinson's Disease. Front Neurol. 2021 Oct 8;12:688760. doi: 10.3389/fneur.2021.688760. eCollection 2021. PMID 34690908
- [Background] Okun MS. Deep-brain stimulation for Parkinson's disease. N Engl J Med. 2012 Oct 18;367(16):1529-38. doi: 10.1056/NEJMct1208070. No abstract available. PMID 23075179
- [Background] Chaudhuri KR, Martinez-Martin P, Schapira AH, Stocchi F, Sethi K, Odin P, Brown RG, Koller W, Barone P, MacPhee G, Kelly L, Rabey M, MacMahon D, Thomas S, Ondo W, Rye D, Forbes A, Tluk S, Dhawan V, Bowron A, Williams AJ, Olanow CW. International multicenter pilot study of the first comprehensive self-completed nonmotor symptoms questionnaire for Parkinson's disease: the NMSQuest study. Mov Disord. 2006 Jul;21(7):916-23. doi: 10.1002/mds.20844. PMID 16547944
- [Background] Morris ME, Huxham F, McGinley J, Dodd K, Iansek R. The biomechanics and motor control of gait in Parkinson disease. Clin Biomech (Bristol). 2001 Jul;16(6):459-70. doi: 10.1016/s0268-0033(01)00035-3. PMID 11427288
- [Background] Rawson KS, Creel P, Templin L, Horin AP, Duncan RP, Earhart GM. Freezing of Gait Boot Camp: feasibility, safety and preliminary efficacy of a community-based group intervention. Neurodegener Dis Manag. 2018 Oct;8(5):307-314. doi: 10.2217/nmt-2018-0022. Epub 2018 Sep 18. PMID 30223709
- [Background] Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol. 2011 Aug;10(8):734-44. doi: 10.1016/S1474-4422(11)70143-0. PMID 21777828
- [Background] Moore O, Peretz C, Giladi N. Freezing of gait affects quality of life of peoples with Parkinson's disease beyond its relationships with mobility and gait. Mov Disord. 2007 Nov 15;22(15):2192-5. doi: 10.1002/mds.21659. PMID 17712856
- [Background] Zhang WS, Gao C, Tan YY, Chen SD. Prevalence of freezing of gait in Parkinson's disease: a systematic review and meta-analysis. J Neurol. 2021 Nov;268(11):4138-4150. doi: 10.1007/s00415-021-10685-5. Epub 2021 Jul 8. PMID 34236501
- [Background] Gonzalez MC, Dalen I, Maple-Grodem J, Tysnes OB, Alves G. Parkinson's disease clinical milestones and mortality. NPJ Parkinsons Dis. 2022 May 12;8(1):58. doi: 10.1038/s41531-022-00320-z. PMID 35550520
- [Background] Diem-Zangerl A, Seppi K, Wenning GK, Trinka E, Ransmayr G, Oberaigner W, Poewe W. Mortality in Parkinson's disease: a 20-year follow-up study. Mov Disord. 2009 Apr 30;24(6):819-25. doi: 10.1002/mds.22414. PMID 19224612
- [Background] Guttman M, Slaughter PM, Theriault ME, DeBoer DP, Naylor CD. Parkinsonism in Ontario: increased mortality compared with controls in a large cohort study. Neurology. 2001 Dec 26;57(12):2278-82. doi: 10.1212/wnl.57.12.2278. PMID 11756610
- [Background] Armstrong MJ, Okun MS. Diagnosis and Treatment of Parkinson Disease: A Review. JAMA. 2020 Feb 11;323(6):548-560. doi: 10.1001/jama.2019.22360. PMID 32044947
- [Background] Lang AE, Lozano AM. Parkinson's disease. Second of two parts. N Engl J Med. 1998 Oct 15;339(16):1130-43. doi: 10.1056/NEJM199810153391607. PMID 9770561
- [Background] Dorsey ER, Constantinescu R, Thompson JP, Biglan KM, Holloway RG, Kieburtz K, Marshall FJ, Ravina BM, Schifitto G, Siderowf A, Tanner CM. Projected number of people with Parkinson disease in the most populous nations, 2005 through 2030. Neurology. 2007 Jan 30;68(5):384-6. doi: 10.1212/01.wnl.0000247740.47667.03. Epub 2006 Nov 2. PMID 17082464
- [Background] Tanner CM, Aston DA. Epidemiology of Parkinson's disease and akinetic syndromes. Curr Opin Neurol. 2000 Aug;13(4):427-30. doi: 10.1097/00019052-200008000-00010. PMID 10970060